CLINICAL TRIAL: NCT06095362
Title: Thyroid Cancer and Lymph Node Metastases Detection Using Bevacizumab-IRDye800CW With Molecular Fluorescence Guided Surgery. Thyroid cAncer Surgery With Intraoperative Molecular fluoRescent Imaging to rEduce overtreatmenT and Morbidity
Brief Title: Thyroid Cancer and Central Lymph Node Metastases Detection Using Bevacizumab-IRDye800CW
Acronym: TARGET-beva
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202000846
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Thyroid Carcinoma; Surgery
Keywords: Optical Molecular Imaging; Molecular Fluorescence Guided Surgery
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Drug: Bevacizumab-IRDye800CW

INTERVENTIONS:
Drug: Bevacizumab-IRDye800CW — All patients will receive a dose of Bevacizumab-IRDye800CW, in a dose of 4.5, 10, or 25mg

SUMMARY:
Background: Papillary thyroid cancer (PTC) patients often develop central lymph node metastases (CLNM), which pose a high risk of disease recurrence. The prophylactic central lymph node dissection (PCLND) is controversial, with proponents arguing for it to prevent local recurrence, and opponents objecting to the hypoparathyroidism and nerve damage risk. Currently, no diagnostic tool exists to identify patients who would benefit from a PCLND. Molecular Fluorescence Guided Surgery (MFGS) is a potential solution that uses fluorescent tracers to detect cancerous tissue. This study aims to investigate whether the administration of a GMP-produced near infrared (NIR) tracer, bevacizumab-IRDye800CW, targeting VEGF-A, can enable intraoperative selection of PTC/FTC/HTC patients for CLND.

Objective: The primary objective of the study is to determine the optimal dose of bevacizumab-IRDye800CW for an adequate tumor-to-background ratio (TBR) in PTC/FTC/HTC lymph node metastases. The secondary objectives are to evaluate the feasibility of MFGS for PTC/FTC/HTC and nodal metastasis assessment, to correlate and validate fluorescence signals detected in vivo with ex vivo histopathology and immunohistochemistry, to evaluate the distribution of bevacizumab-IRDye800CW on a microscopic level, and to quantify the sensitivity and specificity of bevacizumab-IRDye800CW for PTC/FTC/HTC and nodal metastasis.

Study Design: The TARGET-BEVA study is a non-randomized, non-blinded, prospective, single-center phase I feasibility study for patients with confirmed PTC/FTC/HTC, for which the best TBR dosage group in PTC/FTC/HTC nodal metastasis will be determined. The study will initiate with a 3 x 3 scheme: 4,5 mg, 10 mg, and 25 mg, with three patients confirmed with lymph node metastasis in each group. Dosages will be based on previous studies, with the primary objective being the detection of lymph node metastasis. After the first 9 patients, an interim analysis will be performed, after which the best dosage group will be expanded with another 7 patients.

Conclusion: The study aims to identify a novel diagnostic tool that can aid clinicians in selecting patients for PCLND, enabling a reduction in overtreatment, morbidity, and costs while maintaining effectiveness with a lower recurrence rate and improved quality of life.

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 18 years, eligible for surgery
2. Bethesda VI fine needle aspiration (FNA) thyroid or FNA proven PTC/FTC/HTC metastasis (primary or recurrence).
3. Scheduled to undergo central and/or lateral lymph node dissection with or without thyroidectomy as discussed in the Multi-Disciplinary Thyroid Board.
4. WHO performance score of 0-2.
5. Written informed consent.
6. Mentally competent person who is able and willing to comply with study procedures.
7. For female subjects who are of childbearing potential are premenopausal with intact reproductive organs or are less than two years post-menopausal:

   * A negative serum pregnancy test prior to receiving the tracer
   * Willing to ensure that she or her partner uses effective contraception during the trial and for 3 months thereafter.

Exclusion criteria

1. Pregnancy or breast feeding
2. Advanced stage thyroid cancer not suitable for surgical resection
3. Medical or psychiatric conditions that compromise the patient's ability to give informed consent
4. Concurrent anticancer therapy (chemotherapy, radiotherapy, vaccines, immunotherapy) delivered within the last three months prior to the start of the treatment
5. The subject has been included previously in this study or has been injected with another investigational medicinal product within the past six months
6. History of myocardial infarction (MI), TIA, CVA, pulmonary embolism, uncontrolled congestive heart failure (CHF), significant liver disease, unstable angina within 6 months prior to enrollment
7. Any significant change in their regular prescription or non-prescription medication between 14 days and 1 day prior to IMP administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Fluorescent signal levels defined as Tumor-to-Background Ratio (TBR) derived from PTC/FTC/HTC nodal metastasis and normal tissue to determine the optimal dose of Bevacizumab-800CW in patients with PTC/FTC/HTC | Whole study

SECONDARY OUTCOMES:
Correlation of the fluorescent signal assessed by MFGS with other biological and molecular parameters (IHC) and the fluorescent signal assessed in the ex vivo biopsy specimens. | through study completion, an average of 2 years
Wound bed biopsy specimen characteristics (number of positive and negative biopsies. | through study completion, an average of 2 years
Distribution of bevacizumab-IRDye800CW in PTC/FTC/HTC, lymph nodes and normal tissue as identified by SDS-PAGE and/or ELISA and/or fluorescence microscopy. | through study completion, an average of 2 years
Quantification of sensitivity and specificity of Bevacizumab-800CW in order to make a power size calculation for a possible subsequent diagnostic accuracy study. | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Optical Molecular Imaging Group Groningen — http://www.omig.nl